ICare Tonometry Effects on Keratometry Readings, Topography Readings, and Corneal Staining IRB Study # 170608-1 P.I. Kenneth A. Beckman, M.D.

## **Testing Protocol**

Following patient identification and informed consent, a technician will perform visual acuity testing, IOL Master testing, and Pentacam topography testing. The investigator will not be provided with the test results until after the exam is completed.

One drop of saline will be placed on a fluorescein strip. The fluorescein will then be applied to each eye in the inferior fornix. The investigator will evaluate corneal staining using the Oxford staining score for each eye.

The technician will than randomly select a study eye with a coin flip. Once the study eye is identified, the technician will perform ICare tonometry in the study eye only. The IOP will be recorded on the study document, but the investigator will not know which eye was tested.

One drop of saline will be placed on a fluorescein strip. The fluorescein will then be applied to each eye in the inferior fornix. The investigator will evaluate corneal staining using the Oxford staining score for each eye.

The technician will perform IOL Master testing and Pentacam topography testing. The investigator will not be provided with the test results until after the exam is completed.

The technician will then perform ICare tonometry testing in the control eye.

The study eye will then be identified to the investigator and recorded on the study document.

The values from the IOL Master and Pentacam will be transcribed from the printouts onto the study document.

Original copies of the IOL Master and Pentacam tests will be included with the study documents.

V.1, 30 August, 2017